CLINICAL TRIAL: NCT00434226
Title: A Randomized, Controlled, Open-Label, Multicenter, Phase II Study of the Safety and Efficacy of Sunitinib in Combination With Bevacizumab, Carboplatin, and Paclitaxel in Previously Untreated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: A Study of Sunitinib in Combination With Bevacizumab, Carboplatin, and Paclitaxel in Patients With Advanced Non-Small Cell Lung Cancer (SABRE-L)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on data collected, the combination appeared to be poorly tolearated.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clincal Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVF3996g
Record Dates: First submitted 2007-02-11; First posted 2007-02-13 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: SABER-L; NSCLC; Avastin; Sutent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Sunitinib; Carboplatin; Paclitaxel

ARMS (2):
- Bevacizumab + Carboplatin/Paclitaxel + Sunitinib (Experimental)
  Interventions: Drug: bevacizumab; Drug: sunitinib; Drug: carboplatin; Drug: paclitaxel
- Bevacizumab + Carboplatin/Paclitaxel (Placebo Comparator)
  Interventions: Drug: bevacizumab; Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: bevacizumab — Intravenously at a dose of 15mg/kg on the first day of each 21-day cycle
Drug: sunitinib — 25 mg/day for 2 weeks, followed by 1 week of rest
  Arms: Bevacizumab + Carboplatin/Paclitaxel + Sunitinib
Drug: carboplatin — On the first day of each cycle for 4 cycles
Drug: paclitaxel — On the first day of each cycle for 4 cycles

SUMMARY:
This is a Phase II, randomized, controlled, open-label, multicenter trial designed to provide a preliminary assessment of the safety and efficacy of sunitinib when combined with carboplatin and paclitaxel chemotherapy and bevacizumab in patients with locally advanced, recurrent or metastatic NSCLC who have not received prior systemic therapy for NSCLC. All patients will have advanced, histologically or cytologically confirmed NSCLC (Stage IIIb with pleural effusions, Stage IV, or recurrent).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* Advanced histologically or cytologically confirmed NSCLC (Stage IIIb with malignant pleural or pericardial effusion, Stage IV, or recurrent)
* Measurable or non-measurable disease
* Patients with treated brain metastases are eligible if there is no evidence of progression or hemorrhage after treatment, as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period (brain imaging to be competed Day -7 to Day 1).
* Prior treatment for CNS disease as deemed appropriate by the treating physician
* ECOG performance status 0 or 1
* Ability and willingness to comply with study and follow-up procedures

Exclusion Criteria:

* Prior systemic chemotherapy for metastatic disease
* Active malignancy other than lung cancer
* Current, recent, or planned participation in another experimental drug study
* Prior treatment with anti-VEGF agent or agents targeting similar pathways as sunitinib
* Adjuvant chemotherapy or prior combined modality neoadjuvant therapy (chemotherapy plus radiotherapy with or without surgery) within 6 months prior to Day 1 of Cycle 1
* Life expectancy of < 12 weeks
* Current, recent, or planned participation in an experimental drug study
* Inability to take oral medication or requirement of IV alimentation or total parenteral nutrition, or prior surgical procedures affecting absorption
* Inadequate organ function
* Known evidence of disseminated intravascular coagulopathy
* Active infection or fever > 38.5°C within 3 days prior to Day 1 of Cycle 1
* Untreated abnormal thyroid function tests as defined by institutional standards (patients with controlled hypothyroidism are eligible for study participation)
* Any other medical condition(s) (including mental illness or substance abuse) deemed by the clinician to be likely to interfere with a patient's ability to provide informed consent, cooperate, or participate in the study, or to interfere with the interpretation of the results
* Intrathoracic lung carcinoma of squamous cell histology
* Known CNS disease except for treated brain metastases
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Class II or greater CHF
* History of myocardial infarction or unstable angina within 12 months prior to Day 1 of Cycle 1
* History of stroke or transient ischemic attack within 12 months prior to Day 1 of Cycle 1
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection) or recent peripheral arterial thrombosis within 6 months prior to Day 1 of Cycle 1
* History of hemoptysis within 1 month prior to Day 1 of Cycle 1
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1 or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to Day 1 of Cycle 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1 of Cycle 1
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Proteinuria at screening, as demonstrated by a urine protein/creatinine ratio of ≥ 1.0 at screening
* Known hypersensitivity to any component of bevacizumab or sunitinib
* Pregnancy (positive pregnancy test) or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hambleton, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Carboplatin/Paclitaxel + Sunitinib: Bevacizumab intravenously at a dose of 15mg/kg on the first day of each 21-day cycle, carboplatin/paclitaxel on the first day of each cycle for 4 cycles, and sunitinib 25 mg/day for 2 weeks, followed by 1 week of rest
- Bevacizumab + Carboplatin/Paclitaxel: Bevacizumab intravenously at a dose of 15mg/kg on the first day of each 21-day cycle and carboplatin/paclitaxel on the first day of each cycle for 4 cycles
Period: Overall Study
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel
Started | 30 | 26
Completed | 0 | 0
Not Completed | 30 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel | Total
Number analyzed (Participants) | 30 | 26 | 56
Age Continuous [Mean (Standard Deviation); unit: years] — Intent-to-treat population
  years | 63.7 (9.5) | 64.8 (10.7) | 64.2 (10.0)
Age, Customized [Number; unit: participants] — Intent-to-treat population
  participants
    <18 Years | 0 | 0 | 0
    Between 18 and 64 Years | 15 | 13 | 28
    >=65 Years | 15 | 13 | 28
Sex: Female, Male [Count of Participants; unit: Participants] — Intent-to-treat population
  Participants
    Female | 14 | 12 | 26
    Male | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Best Response
Description: The best overall response is the best response, per RECIST criteria, recorded from randomization until disease progression/recurrence (includes both confirmed and unconfirmed responses). Although the original primary outcome was progression-free survival, there was insufficient data available to report on that outcome.
Time Frame: From randomization until disease progression/recurrence
Population: Randomized patients with at least one scan available at baseline and post-baseline
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 25 | 19
participants
  Complete Response | 0 | 0
  Partial Response | 12 | 9
  Stable Disease | 10 | 9
  Progressive Disease | 2 | 1
  Unable to Evaluate | 0 | 0
  Missing | 1 | 0

2. Secondary Outcome: Serious Adverse Events
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 60 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 29 | 26
participants
  Anaemia | 0 | 1
  Febrile Neutropenia | 4 | 1
  Neutropenia | 1 | 0
  Thrombocytopenia | 1 | 0
  Cardiac Arrest | 1 | 1
  Diarrhoea | 1 | 0
  Asthenia | 0 | 1
  Disease Progression | 1 | 1
  Fatigue | 1 | 0
  Pain | 0 | 1
  Hepatic Pain | 0 | 1
  Drug Hypersensitivity | 0 | 1
  Cellulitis | 1 | 0
  Bacterial Sepsis | 0 | 1
  Collapse of Lung | 1 | 0
  Platelet Count Decreased | 1 | 0
  Haemoglobin Decreased | 0 | 1
  Nutrophil Count Decreased | 0 | 1
  Dehydration | 2 | 1
  Back Pain | 1 | 0
  Lung Cancer Metastatic | 0 | 2
  Gastric Cancer | 1 | 0
  Non-Small Cell Lung Cancer | 1 | 0
  Confusional State | 0 | 1
  Renal Failure | 0 | 1
  Pleural Effusion | 0 | 2
  Pneumothorax | 1 | 0
  Chronic Obstructive Pulmonary Disease | 0 | 2
  Pulmonary Embolism | 2 | 0
  Dyspnoea | 0 | 1
  Haemoptysis | 0 | 1
  Pneumonitis | 1 | 0
  Pulmonary Haemorrhage | 0 | 1
  Nasal Septum Perforation | 1 | 0
  Aortic Aneurysm | 1 | 0
  Hypotension | 0 | 1

3. Secondary Outcome: Incidence of Grade ≥ 3 Adverse Events
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 60 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 29 | 26
participants
  Anaemia | 1 | 0
  Febrile Nutropenia | 4 | 2
  Leukopenia | 6 | 3
  Neutropenia | 18 | 12
  Thrombocytopenia | 7 | 5
  Cardiac Arrest | 1 | 1
  Left Ventricular Dysfunction | 1 | 0
  Diarrhoea | 1 | 1
  Gastrointestinal Haemorrhage | 1 | 0
  Asthenia | 0 | 1
  Disease Progression | 1 | 1
  Fatigue | 2 | 3
  Pain | 1 | 2
  Hepatic Pain | 0 | 1
  Drug Hypersensitivity | 0 | 1
  Hypersensitivity | 0 | 1
  Bacterial Sepsis | 0 | 1
  Cellulitis | 1 | 0
  Infection | 1 | 0
  Pneumonia | 0 | 2
  Collapse of Lung | 1 | 0
  Aspartate Aminotransferase Increased | 1 | 0
  Blood Alkaline Phosphatase Increased | 1 | 0
  Fibrin D Dimer Increased | 1 | 0
  Haemoglobin Decreased | 0 | 1
  International Normalised Ratio Increased | 1 | 1
  Nutrophil Count Decreased | 1 | 1
  Platelet Count Decreased | 4 | 0
  White Blood Cell Count Decreased | 2 | 0
  Anorexia | 1 | 0
  Dehydration | 2 | 1
  Hyperglycaemia | 0 | 2
  Hypoalbuminaemia | 1 | 0
  Hypocalcaemia | 0 | 1
  Hyponatraemia | 0 | 2
  Arthralgia | 0 | 1
  Back Pain | 1 | 0
  Muscular Weakness | 1 | 0
  Musculoskeletal Pain | 1 | 0
  Gastric Cancer | 1 | 0
  Lung Cancer Metastatic | 0 | 2
  Metastases to Central Nervous System | 1 | 0
  Non-Small Cell Lung Cancer | 1 | 0
  Dizziness | 1 | 0
  Confusional State | 0 | 1
  Albuminuria | 1 | 0
  Renal Failure | 0 | 1
  Chronic Obstructive Pulmonary Disease | 0 | 1
  Dyspnoea | 2 | 2
  Pleural Effusion | 0 | 2
  Pneumonitis | 1 | 0
  Pulmonary Embolism | 2 | 1
  Pulmonary Haemorrhage | 0 | 1
  Leukocytoclastic Vasculitis | 1 | 0
  Rash | 2 | 0
  Aortic Aneurysm | 1 | 0
  Hypertension | 3 | 1

4. Secondary Outcome: Incidence of Adverse Events Leading to Sunitinib Discontinuation, Dose Interruption, or Dose Reduction
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 60 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib
Number analyzed (Participants) | 29
participants
  Anaemia | 1
  Febrile Nutropenia | 2
  Leukopenia | 4
  Neutropenia | 11
  Thrombocytopenia | 6
  Left Ventricular Dysfunction | 1
  Diarrhoea | 1
  Gastrointestinal Haemorrhage | 1
  Nausea | 1
  Stomatitis | 1
  Disease Progression | 1
  Fatigue | 2
  Bronchitis | 1
  Cellulitis | 1
  Infection | 1
  Collapse of Lung | 1
  Aspartate Aminotransferase Increased | 1
  Fibrin D Dimer Increased | 1
  International Normalised Ratio Increased | 1
  Neutrophil Count Decreased | 1
  Platelet Count Decreased | 5
  White Blood Cell Count Decreased | 1
  Anorexia | 1
  Dehydration | 2
  Hypoalbuminaemia | 1
  Back Pain | 1
  Muscular Weakness | 1
  Musculoskeletal Pain | 1
  Gastric Cancer | 1
  Metastases to Central Nervous System | 1
  Non-Small Cell Lung Cancer | 1
  Dizziness | 1
  Albuminuria | 1
  Pnemothorax | 1
  Dyspnoea | 2
  Pulmonary Embolism | 2
  Leukocytoclastic Vasculitis | 1
  Rash | 1
  Aortic Aneurysm | 1
  Hypertension | 3

5. Secondary Outcome: Incidence of Adverse Events Leading to Bevacizumab Discontinuation or Dose Interruption
Description: All grades according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), v3.0
Time Frame: 60 days following the last administration of study treatment
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Bevacizumab + Carboplatin/Paclitaxel + Sunitinib | Bevacizumab + Carboplatin/Paclitaxel
Number analyzed (Participants) | 29 | 26
participants
  Anaemia | 1 | 0
  Febrile Nutropenia | 1 | 1
  Leukopenia | 1 | 1
  Neutropenia | 3 | 1
  Thrombocytopenia | 3 | 2
  Cardiac Arrest | 0 | 1
  Diarrhoea | 1 | 0
  Gastrointestinal Haemorrhage | 1 | 0
  Disease Progression | 1 | 2
  Fatigue | 2 | 1
  Drug Hypersensitivity | 0 | 1
  Hypersensitivity | 0 | 1
  Bronchitis | 1 | 0
  Infection | 1 | 0
  Collapse of Lung | 1 | 0
  Aspartate Aminotransferase Increased | 1 | 0
  International Normalised Ratio Increased | 1 | 0
  Neutrophil Count Decreased | 0 | 1
  Platelet Count Decreased | 5 | 0
  Dehydration | 2 | 0
  Back Pain | 1 | 0
  Gastric Cancer | 1 | 0
  Lung Cancer Metastatic | 0 | 1
  Metastases to Central Nervous System | 1 | 0
  Metastases to Liver | 0 | 1
  Non-Small Cell Lung Cancer | 1 | 0
  Albuminuria | 1 | 0
  Renal Failure | 0 | 1
  Haemoptysis | 0 | 1
  Pleural Effusion | 0 | 1
  Pneumothorax | 1 | 0
  Pulmonary Embolism | 2 | 0
  Rash | 1 | 0
  Aortic Aneurysm | 1 | 0
  Hypertension | 2 | 2
  Hypotension | 0 | 1

LIMITATIONS AND CAVEATS:
Based on the early safety results from this study, Genentech halted further recruitment and discontinued treatment. Insufficient efficacy data was available to perform additional analyses and limited the interpretation of the analyses performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study.